CLINICAL TRIAL: NCT06442579
Title: The Influence of Cortical Lateralization on Selective Motor Control of the Arm Swing During Independent Walking After Stroke.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); VU University of Amsterdam (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ONZ-2024-0089; 11PEU24N (Other Grant/Funding Number: FWO)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Stroke
Keywords: EMG; EEG; Gait; Arm swing; Kinematics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke (Experimental): Persons with a unilateral first ever stroke
  Interventions: Other: Walking on a treadmill
- Control (Active Comparator): Age and gender matched healthy controls
  Interventions: Other: Walking on a treadmill

INTERVENTIONS:
Other: Walking on a treadmill — Participants have to walk without holding handrails and without bodyweight support for at least 200 gait cycles. They are asked to walk at comfortable walking speed while watching forward to a screen without virtual reality projection. Arm should be next to the body to allow arm swing if possible.

SUMMARY:
The upper limbs play an essential role for safe and efficient walking in healthy persons and persons post-stroke. Nevertheless, in current post-stroke gait rehabilitation (research) the upper limbs are barely targeted. To address this gap, my project aims to investigate the selective motor control of the upper limbs during walking and the contribution of the cortical activity to the arm swing in independent walkers after stroke.

To gain insight in the direct effects of stroke on the arm swing, the primary motor control of the arm swing will be evaluated by determining muscle synergies (i.e group of muscles working together as a task-specific functional unit). Additionally, the cortical activity (EEG-analysis) during walking of persons post-stroke will be compared to healthy controls and the relationship between stroke-induced changes in cortical activity and arm swing deviations will be assessed. Furthermore, I will evaluate whether improvements in cortical activity relate to improvements in primary motor control of the arm swing.

This innovative project will be the first to investigate the direct coupling between the cortex and the muscle synergies in persons post-stroke during independent walking to investigate the arm swing. These fundamental insights in the primary motor control of the arm swing and the contribution of the cortical activity will allow to develop targeted interventions aiming to improve arm swing and as such optimize post-stroke gait rehabilitation.

Research questions:

1. How can muscle synergies explain arm swing alterations in independent walkers after stroke?
2. How do stroke-induced changes in cortical activity relate to arm swing deviations in persons after stroke?
3. Are changes in primary motor control of the upper limb during walking related to normalization of brain activity in independent walkers after stroke?

ELIGIBILITY:
Stroke

Inclusion Criteria:

* First-ever and cerebral stroke
* Able to walk at least 10 minutes (FAC ≥ 3)
* Presence of upper limb paresis (NIHSS item 5a/b > 0)

Exclusion Criteria:

* Other neurological disorders

Healthy controls

Inclusion criteria:

* Older than 18 years
* Able to walk at least 10 minutes

Exlusion criteria:

* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of muscle synergies | Single point of assessment at inclusion
  The number of muscle synergies needed to account for 90% variance in muscle activity measured by surface EMG during walking in stroke survivors compared to healthy controls. Following muscles will be examined:
  * tibialis anterior,
  * gastrocnemius lateralis
  * soleus
  * vastus medialis
  * vastus lateralis
  * rectus femoris
  * biceps femoris
  * gluteus medius
  * erector spinae
  * latissimus dorsi
  * anterior deltoid
  * posterior deltoid
  * biceps brachii
  * triceps brachii
Number of muscle synergies | Single point of assessment 3 months after inclusion (only for stroke survivors)
  The number of muscle synergies needed to account for 90% variance in muscle activity measured by surface EMG during walking in stroke survivors after a follow-up period of three months. Following muscles will be examined:
  * tibialis anterior,
  * gastrocnemius lateralis
  * soleus
  * vastus medialis
  * vastus lateralis
  * rectus femoris
  * biceps femoris
  * gluteus medius
  * erector spinae
  * latissimus dorsi
  * anterior deltoid
  * posterior deltoid
  * biceps brachii
  * triceps brachii
Weight of muscle synergies | Single point of assessment at inclusion
  The number or distribution of muscle weightings within a synergy during walking in stroke survivors compared to healthy controls.
  The distribution of muscle activation averages over one gait cycle measured by surface EMG of following muscles:
  * tibialis anterior,
  * gastrocnemius lateralis
  * soleus
  * vastus medialis
  * vastus lateralis
  * rectus femoris
  * biceps femoris
  * gluteus medius
  * erector spinae
  * latissimus dorsi
  * anterior deltoid
  * posterior deltoid
  * biceps brachii
  * triceps brachii
Weight of muscle synergies | Single point of assessment 3 months after inclusion (only for stroke survivors)
  The number or distribution of muscle weightings within a synergy during walking in stroke survivors after a follow-up period of three months.
  The distribution of muscle activation averages over one gait cycle measured by surface EMG of following muscles:
  * tibialis anterior,
  * gastrocnemius lateralis
  * soleus
  * vastus medialis
  * vastus lateralis
  * rectus femoris
  * biceps femoris
  * gluteus medius
  * erector spinae
  * latissimus dorsi
  * anterior deltoid
  * posterior deltoid
  * biceps brachii
  * triceps brachii
Brain symmetry index (BSI) | Single point of assessment at inclusion
  The amount of cortical lateralization during walking in stroke survivors compared to healthy controls. The score ranges from -1 to +1 with BSI = 0 reprenting perfect symmetry. Positive values represent higher power in the right hemishere compared to the left hemisphere, vice versa for negative values. For left side lesions, BSI was multiplied by -1.
Brain symmetry index (BSI) | Single point of assessment 3 months after inclusion (only for stroke survivors)
  The amount of cortical lateralization during walking in stroke survivors after a follow-up period of three months. The score ranges from -1 to +1 with BSI = 0 reprenting perfect symmetry. Positive values represent higher power in the right hemishere compared to the left hemisphere, vice versa for negative values. For left side lesions, BSI was multiplied by -1.

SECONDARY OUTCOMES:
Upper limb kinematics | Single point of assessment at inclusion
  Movements of the upper limb during walking measured by 3D kinematics and expressed as angles (°)
Upper limb kinematics | Single point of assessment 3 months after inclusion (only for stroke survivors)
  Movements of the upper limb during walking measured by 3D kinematics and expressed as angles (°)
Cortico-synergy coherence | Single point of assessment at inclusion
  The amount of coherence (i.e. phase locking) between the muscle synergies and cortical activity during walking in stroke survivors compared to healthy controls. Higher values (0-1) indicate a better linear association.
Cortico-synergy coherence | Single point of assessment 3 months after inclusion (only for stroke survivors)
  The amount of coherence (i.e phase locking) between the muscle synergies and cortical activity during walking in stroke survivors after a follow-up period of three months. Higher values (0-1) indicate a better linear association.

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | Single point of assessment at inclusion (only for stroke survivors)
  Quantifies the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The highest score is 42.
National Institutes of Health Stroke Scale (NIHSS) | Single point of assessment 3 months after inclusion (only for stroke survivors)
  Quantifies the general impairment caused by a stroke after a follow-up period of three months. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The highest score is 42.
Fugl-Meyer assesment - Upper limbs | Single point of assessment at inclusion (only for stroke survivors)
  Assesses specifc motor impairments of the upper limbs of stroke survivors. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. However, reflex activity is measured using 2 points only, with a score of 0 or 2 for absence and presence of reflex respectively.
Fugl-Meyer assesment - Upper limbs | Single point of assessment 3 months after inclusion (only for stroke survivors)
  Assesses specifc motor impairments of the upper limbs of stroke survivors after a follow-up period of three months. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. However, reflex activity is measured using 2 points only, with a score of 0 or 2 for absence and presence of reflex respectively.
Tardieu scale | Single point of assessment at inclusion (only for stroke survivors)
  Quantifies spasticity by assessing the muscle's response (0-5) to different stretch velocities (V1, V2 or V3) and by determining the spasticity angle (R1 or R2).
Tardieu scale | Single point of assessment 3 months after inclusion (only for stroke survivors)
  Quantifies spasticity by assessing the muscle's response (0-5) to different stretch velocities (V1, V2 or V3) and by determining the spasticity angle (R1 or R2).
10 Meter Walking Test | Single point of assessment at inclusion (only for stroke survivors)
  Examins the walking capacity of a stroke survivor by measuring how long it takes to walk a distance of 10 meters (in seconds).
10 Meter Walking Test | Single point of assessment 3 months after inclusion (only for stroke survivors)
  Examins the walking capacity of a stroke survivor by measuring how long it takes to walk a distance of 10 meters (in seconds).
Fugl-Meyer assesment - Lower limbs | Single point of assessment at inclusion (only for stroke survivors)
  Assesses specifc motor impairments of the lower limbs of stroke survivors. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. However, reflex activity is measured using 2 points only, with a score of 0 or 2 for absence and presence of reflex respectively.
Fugl-Meyer assesment - Lower limbs | Single point of assessment 3 months after inclusion (only for stroke survivors)
  Assesses specifc motor impairments of the lower limbs of stroke survivors after a follow-up period of three months. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. However, reflex activity is measured using 2 points only, with a score of 0 or 2 for absence and presence of reflex respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Van Bladel, PhD, Principal Investigator — Ghent University and Ghent University Hospital
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium